CLINICAL TRIAL: NCT04459442
Title: Placental Transfusion in the 'Natural' Vaginal Delivery at Term: Effect of Early and Late Umbilical Cord Clamping
Brief Title: Placental Transfusion in the 'Natural' Delivery: Effect of Early and Late Umbilical Cord Clamping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Policlinico Abano Terme (Other)
Responsible Party: Principal Investigator, Vincenzo Zanardo, Professor, Policlinico Abano Terme
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 3278/AT/14
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Hematocrit Anemia; Acidosis
Keywords: Placental transfusion; Natural, two-step delivery; Early cord clamping; Delayed cord clamping
MeSH Terms: conditions — Acidosis; Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Parallel Assignment The investigators conducted a randomized controlled trial (parallel group study with 1:1 randomization), comparing early cord clamping (at 60 seconds) and delayed cord clamping (at 180 seconds) in 90 cases of 'normal', two-step vaginal births.
Who Masked: Investigator
Masking Description: None (Open Label)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early cord clamping (Experimental): Cord clamping at 60 seconds after birth.
  Interventions: Procedure: Umbilical cord clamping at birth.
- Delayed cord clamping (Experimental): Cord clamping at 180 seconds after birth.
  Interventions: Procedure: Umbilical cord clamping at birth.

INTERVENTIONS:
Procedure: Umbilical cord clamping at birth. — Umbilical cord clamping after delivery.
  Other Names: Cord clamping

SUMMARY:
The investigators conducted a randomized controlled trial (parallel group study with 1:1 randomisation) comparing early cord clamping (ECC, at 60 seconds) and delayed cord clamping (DCC, at 180 seconds) in 90 cases of 'normal', two-step vaginal deliveries. DCC may result in a higher blood volume in the newborn, facilitating the maternal-placental-fetal exchange of circulating compounds, without potentially detrimental acidosis.

DETAILED DESCRIPTION:
Introduction: Placental transfusion supports an important blood transfer to the neonate, promoting a more stable transition from fetal to extrauterine life, with the potential to prevent iron deficiency in young children. Several studies have demonstrated that cord clamping timing is greatly relevant for facilitate placental transfusion, the transfer of extra blood from the placenta to the infant in the third stage of labor. Therefore, during' natural', 'two-step delivery umbilical cord management may play a relevant role on blood passage to the neonate and it may affect neonatal hematological values (placental transfusion). The most effective way to manage umbilical cord in in 'natural', two-step delivery remains to be established. Objective: The aim of the present study is to evaluate the effect of two different methods of umbilical cord management ECC vs. DCC) on the placental transfusion, defined by Δ haematocrit (Hct) from arterial cord blood at birth and capillary blood at 48 h of age, accounting for physiological body weight decrease. Secondary outcome included contemporary estimate of pH in arterial cord blood gas analysis at birth.

Material and methods: This is a randomized clinical trial on the effect of different cord management in newborns by 'natural', two-step delivery. After obtaining parental consent, all mothers > 38 weeks' gestation will be assigned to either ECC or DCC group in a 1:1 ratio, according to a randomized sequence generated by an opened, sealed, numbered, opaque envelope containing the cord clamping interventions allocation, ECC (at 1 minute) or DCC (at 3 minutes after delivery).

ELIGIBILITY:
Inclusion Criteria:

Vaginal delivery

Exclusion Criteria:

Cesarean delivery

Ages: 1 Minute to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Placental transfusion. | Second day of life
  Placental transfusion defined by delta hematocrit (Htc) from arterial cord blood at birth and capillaryblood at 48 h of age.
Cord blood pH | Second day of life.
  pH estimate in arterial cord blood gas analysis

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Policlinico Abano Terme, Abano Terme, Padua
  - Policlinico Abano Terme, Abano Terme
  - Padua University Hospital, Padua

IPD SHARING:
Plan to Share IPD: No
No. There is not a plan to make IPD available